CLINICAL TRIAL: NCT05523921
Title: Intrafamilial Transmission of Hepatitis B Virus: Frequency, Risk Factors, and Role of Hepatitis B Vaccination
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Faik Hamed Ahmed, Mohamed Faik Hamed Ahmed, Assiut University
Other Study IDs: Transmission of HBV
Record Dates: First submitted 2022-08-29; First posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: HBV Transmission
Keywords: Intrafamilial transmission of HBV.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of the study is to accomplish two major tasks: the first is to determine the frequency of intra-familial transmission of HBV; the second is trying to explore the potential risk factors of such a transmission .As a secondary aim, immunologic status of the household contacts vaccinated for hepatitis B will be evaluated to assess the efficacy of hepatitis B vaccination and its role in prevention of intra-familial transmission of HBV

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) infection is a global health issue; it is estimated that 257 million persons have chronic HBV (Asgeir et al., 2021). The major routes of HBV transmission include blood, sexual contact, vertical (from infected mothers to her children) and horizontal (between the spouses or children) transmission (Şükran et al., (2018). The household transmission of HBV is also a major health issue; it represents a challenge to the health system. Higher rates of HBV infection were reported among the household contacts of chronic HBV carriers; the prevalence of HBV infection among the family members of patients with chronic HBV can reach to 57%. Factors affecting the risk of transmission include socio-demographic status, family role (infected mothers increase the risk of transmission) and viral markers of the index case (Masomeh et al., 2016).The diagnosis of HBV infection is generally based on serological (hepatitis B surface antigen) and molecular assays (hepatitis B virus deoxyribonucleic acid) (Chen et al., 2017).Although the three-dose vaccination for hepatitis B provides more than 90% seroprotection rates (Van Den Ende C, et al, 2017); approximately 10% of vaccinated persons may be at risk of getting infected.

Available data about the current status of intra-familial transmission of HBV among our community members are lacking; we need to determine the magnitude of such a major public health problem

ELIGIBILITY:
Inclusion Criteria:

* : The household contacts of patients with chronic HBV infection will be included in the study.

Exclusion Criteria:

* Those with prior diagnosis of HBV infection following the date of the primary case infection.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We will provide clinical evaluation, laboratory investigations, and abdominal ultrasonography for every participant of the study. Clinical evaluation will include a detailed questionnaire concerning the potential risk factors of intra-familial transmission of HBV; it will include the kind of family relationship, demographic data, history of hepatitis B vaccination, and the potential routes of HBV transmission. The battery of laboratory work will include hepatitis B surface antigen (for diagnosis of infection), and titer of antibody to hepatitis B surface (for assessment of the immunologic status among non-infected subjects). In addition, liver chemistry panel will be performed for infected patients to help in the assessment of liver disease severity.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Determine the frequency of intra-familial transmission of HBV; & trying to explore the potential risk factors of such a transmission. | Baseline.
  Determine the frequency of intra-familial transmission of HBV; & trying to explore the potential risk factors of such a transmission.

SECONDARY OUTCOMES:
To assess the efficacy of hepatitis B vaccination and its role in prevention of intra-familial transmission of HBV. | Baseline.
  To assess the efficacy of hepatitis B vaccination and its role in prevention of intra-familial transmission of HBV.

REFERENCES:
- See also: .Asgeir J, Bitsatab M, Hailemichael D et al., (2021). Mother-to-Child Transmission of Hepatitis B Virus in Ethiopia. Vaccines, 9, 430. — https://pubmed.ncbi.nlm.nih.gov/33925930/
- See also: Chen E-Q, Feng S, Wang M, Liang L, Zhou L et al., (2017). Serum hepatitis B core-related antigen is a satisfactory surrogate marker of intrahepatic covalently closed circular DNA in chronic hepatitis B. Sci Rep; 7:173. — http://www.nature.com/articles/s41598-017-00111-0
- See also: Masomeh S, Mohammad B, Masoomeh Z et al., (2016). Intra-familial Transmission of Hepatitis B Virus Infection in Arak, Central Iran. Iran J Pathol; 11(4): 328 - 333 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5563930/
- See also: Pournik O, Alavian S, Ghalichi L et al., (2013). Lower intrafamilial transmission rate of hepatitis B in patients with hepatitis d coinfection: a data-miningapproach. Hepat; 13(5). — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3732666
- See also: Şükran K (2018). Laboratory Diagnosis of HBV Viral Hepatitis: Chronic Hepatitis B. p 51-64 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2095015/
- See also: Van Den Ende C, et al. The immunogenicity and safety of GSK's recombinant hepatitis B vaccine in adults: a systematic review of 30 years of experience. Expert Rev Vaccines. 2017 16(8):811-832. — https://pubmed.ncbi.nlm.nih.gov/28573913/